CLINICAL TRIAL: NCT01552642
Title: An Interactive Web-based Intervention to Achieve Healthy Weight in Young Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HD068783
Record Dates: First submitted 2012-03-08; First posted 2012-03-13 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Child; Obesity; Overweight
Keywords: Comprehensive Health Enhancement Support System (CHESS)
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Active Comparator): Intervention Group
  Interventions: Behavioral: face-to-face meetings and access to a website
- Control Group (No Intervention): Control Group

INTERVENTIONS:
Behavioral: face-to-face meetings and access to a website — The intervention group will have 6 weekly face-to-face meetings and will have access to a website.
  Arms: Intervention Group

SUMMARY:
The overall purpose of this study is to develop and implement an effective intervention program designed to prevent and treat obesity in young children.

DETAILED DESCRIPTION:
Study procedures and interventions:

Pre-intervention: a full-day training will occur with a physician and nurse from each clinic site to be trained as "champions" in counseling.

Intervention:

A letter of introduction will be mailed to potential subjects whose child was seen in the last 6 months for a well-child exam whose BMI is greater than or equal to the 85th percentile. After informed consent is obtained, the subjects will be randomized to the intervention or control group. One parent may join the study.

Groups of 10 to 12 parents of overweight and obese 3 to 6 year olds will meet once weekly for 6 weeks at 5:30 to 6:30 pm with the "nurse champion" in the primary care office. Topics to be presented and discussed include authoritative parenting, using the food plan "Go, Slow, and Whoa", increasing physical activity, and behavior change strategies. Sessions will be audiotaped and independently audited to confirm program fidelity. Parenting skills will be discussed at every session.

The intervention group will have access to a website. This site will include information services (instant library with health topics related to nutrition and physical activity and answers to frequently asked questions), web links to other pre-screened sources of information on nutrition and physical activity, local resources for current activities for children and families, personal stories (emphasizing authoritative parenting), interactive discussion group and Ask the Expert (questions will be answered within 48 hours and usually sooner).

ELIGIBILITY:
Inclusion Criteria:

* one parent of a 3-6 year old child with a BMI greater than or equal to the 85th percentile
* Internet access
* English speaking

Exclusion Criteria:

* Children with a developmental disorder
* Children with a chronic underlying disease that may contribute to obesity
* Children taking medication that may interfere with a healthy weight

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2013-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Feasibility | 1 year
  To assess the feasibility of an intervention combining 6 'in-person' group counseling sessions with a 1-year longitudinal web-based component to help parents of overweight children promote healthy behavior change.
Efficacy | 1 year
  To assess the effectiveness of this intervention program to assist parents of overweight and obese 3-6 year olds in promoting: (a) a modest reduction of child BMI-z scores, (b) healthy behavior changes (related to nutrition and physical activity) for their children, and (c) improved parenting skills.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen R Wald, MD, Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - UW East Towne Clinic, Madison, Wisconsin
  - UW Pediatrics at 20 S. Park St, Madison, Wisconsin
  - UW Health West Towne Pediatrics, Madison, Wisconsin

REFERENCES:
- [Background] Spivack JG, Swietlik M, Alessandrini E, Faith MS. Primary care providers' knowledge, practices, and perceived barriers to the treatment and prevention of childhood obesity. Obesity (Silver Spring). 2010 Jul;18(7):1341-7. doi: 10.1038/oby.2009.410. Epub 2009 Nov 12. PMID 19910934
- [Background] Golan M, Weizman A, Apter A, Fainaru M. Parents as the exclusive agents of change in the treatment of childhood obesity. Am J Clin Nutr. 1998 Jun;67(6):1130-5. doi: 10.1093/ajcn/67.6.1130. PMID 9625084
- [Background] Ewing LJ, Cluss P, Goldstrohm S, Ulrich R, Colborn K, Cipriani L, Wald ER. Translating an evidence-based intervention for pediatric overweight to a primary care setting. Clin Pediatr (Phila). 2009 May;48(4):397-403. doi: 10.1177/0009922808330109. Epub 2009 Jan 21. PMID 19164134
- [Background] Wachs JE. Strategies to develop "interconnectedness". Part II Connection within the community. AAOHN J. 1992 Mar;40(3):144-6. No abstract available. PMID 1550624
- [Background] Shaw BR, McTavish F, Hawkins R, Gustafson DH, Pingree S. Experiences of women with breast cancer: exchanging social support over the CHESS computer network. J Health Commun. 2000 Apr-Jun;5(2):135-59. doi: 10.1080/108107300406866. PMID 11010346
- [Background] Gustafson DH, McTavish FM, Boberg E, Owens BH, Sherbeck C, Wise M, Pingree S, Hawkins RP. Empowering patients using computer based health support systems. Qual Health Care. 1999 Mar;8(1):49-56. doi: 10.1136/qshc.8.1.49. No abstract available. PMID 10557670
- [Background] Subar AF, Crafts J, Zimmerman TP, Wilson M, Mittl B, Islam NG, McNutt S, Potischman N, Buday R, Hull SG, Baranowski T, Guenther PM, Willis G, Tapia R, Thompson FE. Assessment of the accuracy of portion size reports using computer-based food photographs aids in the development of an automated self-administered 24-hour recall. J Am Diet Assoc. 2010 Jan;110(1):55-64. doi: 10.1016/j.jada.2009.10.007. PMID 20102828
- [Background] Vartanian VE, Bublik VG. [Late results of correction of flatfoot in children using an electro-myostimulation method]. Ortop Travmatol Protez. 1989 Feb;(2):26-9. Russian. PMID 2786178
- [Result] Savoye M, Shaw M, Dziura J, Tamborlane WV, Rose P, Guandalini C, Goldberg-Gell R, Burgert TS, Cali AM, Weiss R, Caprio S. Effects of a weight management program on body composition and metabolic parameters in overweight children: a randomized controlled trial. JAMA. 2007 Jun 27;297(24):2697-704. doi: 10.1001/jama.297.24.2697. PMID 17595270
- [Result] Golley RK, Magarey AM, Baur LA, Steinbeck KS, Daniels LA. Twelve-month effectiveness of a parent-led, family-focused weight-management program for prepubertal children: a randomized, controlled trial. Pediatrics. 2007 Mar;119(3):517-25. doi: 10.1542/peds.2006-1746. PMID 17332205
- [Result] Wald ER, Moyer SC, Eickhoff J, Ewing LJ. Treating childhood obesity in primary care. Clin Pediatr (Phila). 2011 Nov;50(11):1010-7. doi: 10.1177/0009922811410871. Epub 2011 Jun 6. PMID 21646253